CLINICAL TRIAL: NCT00305669
Title: A Pilot Study of Two Dose Schedules of Granulocyte Macrophage Colony-Stimulating Factor (GM-CSF) as Neo-Adjuvant Therapy in Patients With Localized Prostate Cancer
Brief Title: GM-CSF Before Surgery in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000455649; UCSF-04558; UCSF-H40568-25161-02B
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim; Immunohistochemistry; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-CSF before surgery (Experimental): GM-CSF dose prior to surgery- Cohort 1-GM-CSF 250mcg/m2 for 2 weeks Cohort 2-GM-CSF 250mcg/m2 for 3 weeks Cohort 3-GM-CSF 250mcg/m2 for 4 weeks Cohort 4-GM-CSF 125mcg/m2 for 4 weeks
  Interventions: Biological: sargramostim; Other: immunohistochemistry staining method; Other: immunological diagnostic method; Other: laboratory biomarker analysis; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: sargramostim
Other: immunohistochemistry staining method
Other: immunological diagnostic method
Other: laboratory biomarker analysis
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Colony-stimulating factors, such as GM-CSF, may help the body build an effective immune response to kill tumor cells. Giving GM-CSF before surgery may be an effective treatment for localized prostate cancer.

PURPOSE: This clinical trial is studying how well giving GM-CSF before surgery works in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of daily neoadjuvant sargramostim (GM-CSF) in patients with localized prostate cancer undergoing radical prostatectomy.
* Determine whether tissue-specific antiprostate cancer immunity is induced by the administration of neoadjuvant GM-CSF in patients with localized prostate cancer prior to radical prostatectomy.

Secondary

* Estimate the baseline antitumor immune response in patients treated with 2 different dose schedules of GM-CSF.
* Determine the magnitude of the difference in immune response between 2 dose schedules of GM-CSF.
* Determine the clinical effects, including prostate-specific antigen (PSA) decline, surgical outcome, surgical complications, and histologic appearance of surgical specimen, of this regimen in these patients.

OUTLINE: This is a pilot study. Patients are stratified according to sargramostim (GM-CSF) dose.

Patients receive 1 of 2 dose levels of GM-CSF subcutaneously on days 1-14 or 1-21. Treatment continues in the absence of unacceptable toxicity. Within 3 days after the last dose of GM-CSF, patients undergo radical prostatectomy.

Blood is collected at baseline, day 28 of each course, and at the 4-week follow-up visit and is examined for activated T-cells. Tissue is collected during surgery and assessed for biomarkers and cytokines.

After completion of study treatment, patients are followed at 4 weeks.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate

  * No neuroendocrine or small cell features
* No evidence of metastatic disease
* Planning radical prostatectomy at least 2 months from now
* Testosterone level normal

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 or Karnofsky PS 70-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8 g/dL
* AST and ALT ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* PT and PTT normal
* Fertile patients must use effective barrier contraception
* No history of allergic reaction to compounds of similar chemical or biologic composition to sargramostim (GM-CSF)
* No ongoing or active bacterial, viral, or fungal infection
* DLCO > 50% if patient has a history of clinically significant obstructive airway disease
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No other active malignancy, defined as cancer for which therapy has been completed and patient is now considered < 30% risk of relapse, except nonmelanoma skin cancer
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No underlying medical condition that, in the opinion of the principal investigator, may make the administration of GM-CSF hazardous or obscure the interpretation of adverse events

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior major surgery
* No prior radiotherapy, immunotherapy, chemotherapy, or other investigational therapy for this cancer
* No prior hormonal therapy including any of the following:

  * Luteinizing-hormone releasing hormone (LHRH) agonists
  * LHRH antagonists
  * Antiandrogens, including any of the following:

    * Bilcalutamide
    * Flutamide
    * Nilutamide
  * 5-alpha-reductase inhibitors
  * PC-SPES or other PC-x product
  * Estrogen-containing nutriceuticals
* No concurrent chemotherapy or radiotherapy
* No concurrent systemic steroid therapy

  * Concurrent inhaled or topical steroids allowed
* No other concurrent immunotherapy
* No other concurrent investigational agent
* No other concurrent anticancer agents or therapies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of daily neoadjuvant sargramostim (GM-CSF) in patients with localized prostate cancer undergoing radical prostatectomy. | up to 6 weeks following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Fong, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States